CLINICAL TRIAL: NCT03936244
Title: Randomized Controlled Trial Comparing Bipolar Plasmakinetic Transurethral Resection of the Prostate With Monopolar Transurethral Resection of the Prostate in the Treatment of Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Brief Title: Bipolar Plasmakinetic TURP Vs Monopolar TURP in the Treatment of Lower Urinary Tract Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Fuenlabrada (Other)
Responsible Party: Principal Investigator, Carolina Alonso, Attending physician, Hospital Universitario de Fuenlabrada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUF
Record Dates: First submitted 2019-04-24; First posted 2019-05-03 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Transurethral Resection of Prostate
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- M-TURP (Active Comparator): The M-TURP procedure requires the use of a resectoscope (Olympus or Storz, 26Ch), camera system and irrigation fluid (Glycine 1.5%, Baxter). The system consists of a generator unit (ForceTriadTM, Medtronic) and a stainless steel loop with an electrical current running through the loop used to cut (120W) prostate tissue and cauterize (80W). Prostate tissue is cut away in small pieces and removed at the end of the procedure using an Ellik evacuator
  Interventions: Device: Transurethral Resection of the Prostate (TURP)
- PK-TURP (Experimental): The PK-TURP procedure requires the use of a resectoscope (Storz, 26Ch), camera system and irrigation fluid (NaCl 0.9%, Baxter). The system consists of a generator unit (PlasmaKineticTM Superpulse de Gyrus, ACMI) and a platinum-iridium superloop with an electrical current running through the loop used to cut (180W) prostate tissue and cauterize (100W). Prostate tissue is cut away in small pieces and removed at the end of the procedure using an Ellik evacuator
  Interventions: Device: Transurethral Resection of the Prostate (TURP)

INTERVENTIONS:
Device: Transurethral Resection of the Prostate (TURP) — Randomized allocation to M-TURP or PK-TURP

SUMMARY:
Randomized controlled trial with one-year follow-up comparing intra, peri and postoperative outcomes for plasmakinetic transurethral resection of prostate (PK-TURP) and monopolar transurethral resection of prostate (M-TURP) in the treatment of LUTS due to BPH in a tertiary-care public institution

DETAILED DESCRIPTION:
The study is a randomized controlled trial with one-year follow-up comparing intra, peri and postoperative outcomes (efficacy, complications and sequelae) for plasmakinetic transurethral resection of prostate (PK-TURP) and monopolar transurethral resection of prostate (M-TURP) in the treatment of LUTS due to BPH in a tertiary-care public institution (Madrid, Spain)

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent voluntarily and will be willing to follow-up
* Prostate volume <80 g
* Meet any conditions (1) Diagnose of LUTS due to refractory to drugs BPH. (2) presenting complications derived from BPH (bladder calculi, recurrent haematuria, recurrent urinary tract infections, acute urinary retention)
* The use of antiplatelet agents or anticoagulant drugs is allowed.

Exclusion Criteria:

* Previous history of pelvic surgery
* Previous history of pelvic radiotherapy
* Previous history of neurogenic bladder dysfunction
* Documented or suspected prostate carcinoma
* Patients with severe cardiopulmonary disease or severe mental disorders
* Poor compliance, and can not be followed up.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Álvarez Ardura, M.D., Principal Investigator — Hospital Universitario de Fuenlabrada; Hugo Otaola Arca, M.D., Ph.D., Principal Investigator — Hospital Universitario de Fuenlabrada; Álvaro Páez Borda, M.D., Ph.D., Study Chair — Hospital Universitario de Fuenlabrada
Locations (1):
- Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahyai SA, Gilling P, Kaplan SA, Kuntz RM, Madersbacher S, Montorsi F, Speakman MJ, Stief CG. Meta-analysis of functional outcomes and complications following transurethral procedures for lower urinary tract symptoms resulting from benign prostatic enlargement. Eur Urol. 2010 Sep;58(3):384-97. doi: 10.1016/j.eururo.2010.06.005. Epub 2010 Jun 11. PMID 20825758
- [Background] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Result] Otaola-Arca H, Alvarez-Ardura M, Molina-Escudero R, Fernandez MI, Paez-Borda A. A prospective randomized study comparing bipolar plasmakinetic transurethral resection of the prostate and monopolar transurethral resection of the prostate for the treatment of Benign Prostatic Hyperplasia: efficacy, sexual function, Quality of Life, and complications. Int Braz J Urol. 2021 Jan-Feb;47(1):131-144. doi: 10.1590/S1677-5538.IBJU.2019.0766. PMID 33047918

RESULTS

PARTICIPANT FLOW:
Groups:
- M-TURP: The M-TURP procedure requires the use of a resectoscope (Olympus or Storz, 26Ch), camera system and irrigation fluid (Glycine al 1.5%, Baxter). The system consists of a generator unit (ForceTriadTM, Medtronic) and a stainless steel loop with an electrical current running through the loop used to cut (120W) prostate tissue and cauterize (80W). Prostate tissue is cut away in small pieces and removed at the end of the procedure using an Ellik evacuator
  Transurethral Resection of the Prostate (TURP): Randomized allocation to M-TURP or PK-TURP
Period: Overall Study
Arm/Group | M-TURP | PK-TURP
Started | 57 | 43
Completed | 45 | 39
Not Completed | 12 | 4
Not completed — Lost to Follow-up | 5 | 1
Not completed — Physician Decision | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M-TURP | PK-TURP | Total
Number analyzed (Participants) | 45 | 39 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (7.2) | 66.2 (7.1) | 65.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 45 | 39 | 84
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (4.2) | 26.8 (4.2) | 27.4 (4.2)
Hypertension [Count of Participants; unit: Participants] | 27 | 18 | 45
Diabetes mellitus [Count of Participants; unit: Participants] | 7 | 6 | 13
Smoker [Count of Participants; unit: Participants] | 7 | 6 | 13
ASA classification [Count of Participants; unit: Participants]
  ASA I | 1 | 1 | 2
  ASA II | 38 | 33 | 71
  ASA III | 6 | 5 | 11
Serum PSA [Mean (Standard Deviation); unit: ng/mL] | 2 (3) | 1.3 (0.9) | 1.7 (2.2)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.9 (0.3) | 0.9 (0.1) | 0.9 (0.3)
Serum sodium [Mean (Standard Deviation); unit: mEq/L] | 140.8 (2.3) | 140.5 (2.5) | 140.7 (2.4)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.7 (1.3) | 15.1 (1.1) | 14.9 (1.2)
IPSS [Mean (Standard Deviation); unit: units on a scale] — IPSS = International Prostate Symptom Score
  Interpretation:
  * Is the sum of the 7 items
  * Scale range: between 0 to 35 units on the scale
  * Higher values represent a worse outcome
  * Subcategories: allows categorizing the lower urinary tract symptoms (LUTS) in three categories
    * 0-7 units on the scale: Mild LUTS
    * 8-19 units on the scale: Moderate LUTS
    * 20-35 units on the scale: Severe LUTS
  units on a scale | 24.7 (6.1) | 23.8 (4.8) | 24.3 (6.1)
QoL score [Mean (Standard Deviation); unit: units on a scale] — QoL = Quality of Life
  Interpretation:
  * Is the value of item 8 of the IPSS questionnaire
  * Scale range: between 0 to 6 units on the scale
  * Higher values represent a worse outcome
  * Subcategories: allows categorizing the QoL in three categories
    * 0-2 units on the scale: Good QoL
    * 3 units on the scale: Intermediate QoL
    * 4-6 units on the scale: poor QoL
  units on a scale | 5.2 (0.8) | 4.8 (1.3) | 5.1 (1.1)
Number of Participants Reporting Sexual Activity in the Last Month [Count of Participants; unit: Participants] — All patients were asked, Did you have sexual activity in the last month?
  Possible answers: yes/no
  Participants | 37 | 28 | 65
IIEF score [Mean (Standard Deviation); unit: units on a scale] — IIEF = International Index of Erectile Function
  Interpretation:
  * Is the sum of the 5 items of the questionnaire
  * Scale range: between 1 to 25 units on the scale
  * Higher values represent a better outcome
  * Subcategories: allows categorizing the erectile function of patients:
    * 22-25 units on the scale: Without erectile dysfunction
    * 17-21 units on the scale: Mild erectile dysfunction
    * 12-16 units on the scale: Mild to moderate erectile dysfunction
    * 8-11 units on the scale: Moderate erectile dysfunction
    * 1-7 units on the scale: Severe erectile dysfunction
  units on a scale | 11.7 (7.1) | 10.5 (7.9) | 11.2 (7.5)
Qmax [Mean (Standard Deviation); unit: mL/s] — Maximum urinary flow rate (mL/s) in free uroflowmetry
  mL/s | 10.9 (5.5) | 9.3 (4) | 10.1 (4.9)
PVRU volume [Mean (Standard Deviation); unit: mL] — PVRU = postvoid residual urine
  Postvoid residual urine in the bladder after urination, measured with transvesical ultrasound
  mL | 60.6 (83.4) | 93.1 (91.1) | 75.9 (88.0)
PV by TRUS [Mean (Standard Deviation); unit: mL] | 38.3 (17.4) | 41.4 (17.1) | 39.7 (17.2)
Stress urinary incontinence [Count of Participants; unit: Participants] | 0 | 0 | 0
Urge urinary incontinence with need for drug use (UUIND) [Count of Participants; unit: Participants] | 1 | 2 | 3
urge Urinary incontinence without the need for drug use (UUIWND) [Count of Participants; unit: Participants] | 13 | 9 | 22
Retrograde ejaculation [Count of Participants; unit: Participants] | 5 | 3 | 8
Dysuria [Count of Participants; unit: Participants] | 5 | 6 | 11
Drugs for hemostasis [Count of Participants; unit: Participants]
  None | 31 | 30 | 61
  Antiaggregants | 12 | 5 | 17
  Anticoagulants | 2 | 4 | 6
Drugs for LUTS [Count of Participants; unit: Participants]
  None | 1 | 1 | 2
  Storage symptoms | 1 | 2 | 3
  Voiding symptoms | 43 | 36 | 79
Indication of surgery [Count of Participants; unit: Participants]
  Drug failure | 35 | 28 | 63
  Acute urinary retention (AUR) | 9 | 10 | 19
  Vesical calculi | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS)
Description: International Prostate Symptom Score (with 7 questions) at 1, 3, 6, and 12 months after surgery.
  Results: the sum of the 7 items will range between 0 to 35 points Interpretation: allows categorizing the lower urinary tract symptoms (LUTS) in 3 categories
  * Mild LUTS: 0-7 points
  * Moderate LUTS: 8-19 points
  * Severe LUTS: 20-35 points
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
points
  1 month | 14.6 (7.4) | 12.7 (7.4)
  3 months | 12.2 (8.2) | 11.3 (7.8)
  6 months | 9.7 (7.7) | 9.4 (5.9)
  12 months | 9.7 (8) | 7.4 (4.7)

2. Primary Outcome: Maximum Urinary Flow Rate (Qmax
Description: Maximum urinary flow rate (mL/s) at 1, 3, 6, and 12 months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
mL/s
  1 months | 17.5 (9) | 18.9 (8.3)
  3 months | 18.2 (8.9) | 16.8 (9)
  6 months | 21 (10.1) | 18.7 (8.1)
  12 months | 21.2 (9.5) | 19.2 (7.2)

3. Primary Outcome: Postvoid Residual Urine (PVRU) Volume
Description: Postvoid residual urine volume (mL) was measured by abdominal ultrasound after urination at 1, 3, 6, and 12 months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
mL
  1 month | 14.2 (28.8) | 13 (22.3)
  3 months | 22.8 (44.9) | 18.2 (26.5)
  6 months | 15.3 (28.9) | 14.7 (25)
  12 months | 14 (28.3) | 8.3 (17.7)

4. Secondary Outcome: Quality of Life (QoL): Bother Score Item of the IPSS Questionnaire
Description: We use the bother score item of the IPSS questionnaire (question 8) at 1, 3, 6, and 12 months after surgery to assess the quality of life (QoL) due to lower urinary tract symptoms (LUTS) Results: will range between 0 to 6 points Interpretation: allows categorizing the QoL in 3 categories
  * Good QoL: 0-2 points
  * Intermediate QoL: 3 points
  * Poor QoL: 4-6points
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
points
  1 month | 3.7 (1.9) | 2.9 (2.1)
  3 months | 2.9 (1.8) | 2.6 (1.9)
  6 months | 2.3 (1.9) | 1.6 (1.6)
  12 months | 2.4 (1.9) | 1.5 (1.2)

5. Secondary Outcome: Number of Participants Reporting Sexual Activity in the Last Month
Description: Measure Description: All patients were asked, Did you have sexual activity in the last month? Possible answers were yes or no.
  Possible answers: yes or no.
  Measurement moment: at 1, 3, 6 and 12 months after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 23 | 22
  3 months | 33 | 28
  6 months | 30 | 29
  12 months | 29 | 30

6. Secondary Outcome: International Index of Erectile Function (IIEF-5)
Description: International Index of Erectile Function (with 5 questions) at 1, 3, 6, and 12 months after surgery.
  Results: the sum of the 5 items will range between 1 to 25 points Interpretation: allows categorizing the erectile function of patients
  * Without erectile dysfunction: 22-25 points
  * Mild erectile dysfunction: 17-21 points
  * Mild to moderate erectile dysfunction: 12-16 points
  * Moderate erectile dysfunction: 8-11 points
  * Severe erectile dysfunction: 1-7 points
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
points
  1 month | 8.5 (7.9) | 9.5 (8)
  3 months | 9.9 (8.2) | 10.7 (8.1)
  6 months | 10.7 (8.5) | 12.4 (8.2)
  12 months | 9.7 (8.6) | 11 (8.1)

7. Secondary Outcome: Prostate Volume (PV)
Description: Prostate volume was measured by transrectal ultrasound at 12 months after surgery
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
mL | 22.3 (13) | 22.5 (12.2)

8. Secondary Outcome: Operative Time
Description: Operative time (min)
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
minutes | 39.7 (14.1) | 47.7 (21.4)

9. Secondary Outcome: Irrigation Volume
Description: Irrigation volume (L)
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: L
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
L | 16 (6.8) | 20.2 (11.8)

10. Secondary Outcome: Change in Plasmatic Sodium in 24 Hours Post-operation
Description: Compared with the baseline, to demonstrate the sodium loss during operation
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
mEq/L | 3.3 (4.1) | 2.2 (3.6)

11. Secondary Outcome: Change in Haemoglobin in 24 Hours Post-operation
Description: Compared with the baseline, to demonstrate the blood loss during operation
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
mg/dL | 0.9 (1.1) | 1 (1.1)

12. Secondary Outcome: Transfusion Rate
Description: Number of participants requiring blood transfusion during, expressed in %
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants | 0 | 0

13. Secondary Outcome: Catheter Duration
Description: Catheter duration (days)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
days | 3.6 (1.4) | 3.5 (0.8)

14. Secondary Outcome: Hospital Stay
Description: Hospital stay (days)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
days | 1.1 (0.4) | 1.1 (0.8)

15. Secondary Outcome: Resected Tissue Weigh
Description: Resected tissue weigh (grams)
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
grams | 12.7 (8.2) | 12.4 (9.9)

16. Secondary Outcome: Resected Tissue Percentage
Description: Compared with the baseline, to demonstrate the % of tissue loss during operation
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: % of resected tissue
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
% of resected tissue | 33.5 (17) | 28.8 (19)

17. Secondary Outcome: Speed Resection
Description: Speed resection (g/min)
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
g/min | 0.9 (0.3) | 0.9 (0.3)

18. Secondary Outcome: Early Reoperation Rate
Description: The ratio of patient who need reoperation because bleeding complications
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants | 2 | 1

19. Secondary Outcome: Late Reoperation Rate
Description: The ratio of patient who need reoperation because residual adenoma or complications
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants | 2 | 1

20. Secondary Outcome: Post-TURP Syndrome Rate
Description: Post-transurethral resection of the prostate syndrome rate was recorded.
Time Frame: Up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants | 1 | 0

21. Secondary Outcome: Clavien Dindo System
Description: It is a system for evaluating surgical complications at 12 months after surgery.
  Clavien I
  * Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions.
  * Acceptable therapeutic regimens are drugs as antiemetics, antipyretics, analgesics, diuretics and electrolytes, and physiotherapy.
  Clavien II
  * Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  * Blood transfusions and total parenteral nutrition are also included
  Clavien III
  - Requiring surgical, endoscopic or radiological intervention
  Clavien IV - Life-threatening complication (including central nervous system complications) requiring intensive care unit management
  Clavien V
  - Death of a patient
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  Clavien I | 2 | 2
  Clavien II | 2 | 2
  Clavien III | 2 | 1
  Clavien IV | 0 | 0
  Clavien V | 0 | 0

22. Secondary Outcome: Bleeding Complications Rate
Description: Register the number of events of haematuria and acute urinary retention by clots
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants | 8 | 7

23. Secondary Outcome: Urinary Tract Infections Rate
Description: Register the number of urinary tract infections at 1, 3, 6, and 12 months after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 5 | 1
  3 months | 0 | 0
  6 months | 0 | 0
  12 months | 0 | 0

24. Secondary Outcome: Stenotic Complications Rate: Meatal Stenosis
Description: Register the number of meatal stenosis at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 2 | 2
  3 months | 5 | 2
  6 months | 2 | 0
  12 months | 4 | 2

25. Secondary Outcome: Stenotic Complications Rate: Urethral Stricture
Description: Register the number of urethral stricture at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 0 | 0
  3 months | 2 | 1
  6 months | 2 | 2
  12 months | 1 | 2

26. Secondary Outcome: Stenotic Complications Rate: Bladder Neck Contracture
Description: Register the number of bladder neck contracture at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 0 | 0
  3 months | 1 | 0
  6 months | 2 | 0
  12 months | 1 | 0

27. Secondary Outcome: Stress Urinary Incontinence Rate
Description: Register the number of patients with stress urinary incontinence at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 18 | 12
  3 months | 12 | 9
  6 months | 7 | 3
  12 months | 3 | 0

28. Secondary Outcome: Urge Urinary Incontinence With Need for Drug Use (UUIND) Rate
Description: Register the number of patients with urge urinary incontinence with need for drug use at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 9 | 3
  3 months | 3 | 3
  6 months | 3 | 2
  12 months | 0 | 0

29. Secondary Outcome: Urge Urinary Incontinence Without Need for Drug Use (UUIWND) Rate
Description: Register the number of patients with urge urinary incontinence without need for drug use at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 8 | 4
  3 months | 6 | 3
  6 months | 6 | 4
  12 months | 1 | 0

30. Secondary Outcome: Sequelae Rate: Retrograde Ejaculation
Description: register the number of retrograde ejaculation at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 17 | 13
  3 months | 24 | 18
  6 months | 21 | 17
  12 months | 23 | 18

31. Secondary Outcome: Sequelae Rate: Dysuria
Description: register the number of dysuria at 1, 3, 6, and 12 after surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | M-TURP | PK-TURP
Number analyzed (Participants) | 45 | 39
Participants
  1 month | 5 | 0
  3 months | 0 | 0
  6 months | 0 | 0
  12 months | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Clavien-Dindo classification
Arm/Group | M-TURP | PK-TURP
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/45 | 1/39
Other Adverse Events (participants affected / at risk) | 4/45 | 4/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M-TURP (N=45) | PK-TURP (N=39)
Need for reintervention (Renal and urinary disorders) | 2 | 1 — Need for surgery because of residual adenoma, urethral stenosis or bladder neck contracture
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-TURP (N=45) | PK-TURP (N=39)
Stenotic events without the need for surgery (Renal and urinary disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03936244/Prot_SAP_000.pdf